CLINICAL TRIAL: NCT03358875
Title: A Phase 3, Open-Label, Multicenter, Randomized Study to Investigate the Efficacy and Safety of BGB-A317 (Anti-PD1 Antibody) Compared With Docetaxel in Patients With Non-Small Cell Lung Cancer Who Have Progressed on a Prior Platinum-Containing Regimen
Brief Title: Comparison of Efficacy and Safety of Tislelizumab (BGB-A317) Versus Docetaxel as Treatment in the Second- or Third-line Setting in Participants With Non-Small Cell Lung Cancer (NSCLC)
Acronym: RATIONALE-303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-303; 2018-000245-39 (EudraCT Number); CTR20171112 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab (Experimental): Participants received tislelizumab 200 mg intravenously (IV) once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of informed consent, whichever occurred first.
  Interventions: Drug: Tislelizumab
- Docetaxel (Active Comparator): Participants received docetaxel 75 mg/m² IV once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of informed consent, whichever occurred first.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab administered by intravenous (IV) infusion
  Other Names: BGB-A317; TEVIMBRA®
  Arms: Tislelizumab
Drug: Docetaxel — Docetaxel administered as an IV infusion over 1 hour
  Arms: Docetaxel

SUMMARY:
The purpose of this study is to show that tislelizumab will improve overall survival in participants with Stage IIIB or IV non-small cell lung cancer when compared to docetaxel in second or third-line treatment setting.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter Phase 3 study in adult participants with histologically confirmed, locally advanced or metastatic (Stage IIIB or IV), NSCLC (squamous or non-squamous) who have disease progression during or after a platinum-containing regimen.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years.
2. Signed Informed Consent Form.
3. Histologically confirmed locally advanced or metastatic (Stage IIIB or IV) NSCLC of either squamous or non-squamous histology types with disease progression during or following treatment with at least one platinum-containing regimen, but no more than 2 lines of systemic therapy.
4. Participants must be able to provide fresh or archival tumor tissues for central assessment of PD-L1 expression in tumor cells. Participants with non-squamous histology must provide evidence of not harboring sensitizing epidermal growth factor (EGFR) mutation tested by a histology-based method.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
6. Adequate hematologic and end-organ function.
7. Expected life span > 12 weeks.
8. Willing to be compliance with birth control requirement during pre-specified study participating period

Key Exclusion Criteria:

1. Prior therapies of docetaxel or treatment targeting programmed cell death protein 1 (PD-1), PD-L1 or cytotoxic T-lymphocyte associated protein 4 (CTLA-4).
2. Harboring EGFR sensitizing mutation or anaplastic lymphoma kinase (ALK) gene translocation.
3. Unresolved side effects of Grade 2 and above from prior anti-cancer therapies, except for adverse events (AEs) not constituting a likely safety risk (e.g. alopecia, rash, pigmentation, specific lab abnormalities).
4. History of severe hypersensitivity reactions to other monoclonal antibodies (mAbs).
5. History of interstitial lung disease, non-infectious pneumonitis or participants with significantly impaired pulmonary function, or who require supplemental oxygen at baseline.
6. With uncontrollable pleural effusion, pericardial effusion, or clinically significant ascites requiring interventional treatment.
7. Active leptomeningeal disease or uncontrolled, untreated brain metastasis.
8. Severe chronic or active infection requiring systemic treatment.
9. Known human immunodeficiency virus (HIV) infection, participants with untreated chronic hepatitis B, active vaccination treatment.
10. Insufficient cardiac functions and other underlying unfavorable cardiovascular conditions.
11. Prior allogeneic stem cell transplantation or organ transplantation.
12. Active autoimmune diseases or history of autoimmune diseases that may relapse.
13. With conditions requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications.
14. With severe underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse that may affect the explanation of drug toxicity or AEs or result in impaired compliance with study conduct.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2024-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (121):
- Brazil (16):
  - Hospital de Amor Barretos, Barretos
  - Hospital Evangelico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim
  - Hospital Haroldo Juacaba Instituto Do Cancer Do Ceara, Fortaleza
  - Oncosite Centro de Pesquisa Clinica Em Oncologia, Ijuí
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Hospital Bruno Born, Lajeado
  - Hospital Sao Vicente de Paulo, Passo Fundo
  - Hgb Hospital Giovanni Battista Mae de Deus Center, Porto Alegre
  - Hospital Sao Lucas Da Pucrs, Porto Alegre
  - Hospital Nossa Senhora Da Conceicao, Porto Alegre
  - Hospital de Clinicas de Porto Alegre, Porto AlegreRS
  - Inca Instituto Nacional de Cancer, Rio de Janeiro
  - Nob Nucleo de Oncologia Da Bahia, Salvador
  - Cepho Centro de Estudos E Pesquisas de Hematologia E Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, São José do Rio Preto
  - Icesp Instituto Do Cancer Do Estado de Sao Paulo Octavio Frias de Oliveira, São Paulo
- Bulgaria (6):
  - Umhat Deva Maria, Eood, Burgas
  - Mhat Dobrich, Ad, Dobrich
  - Mhat Dr Tota Venkova, Ad, Gabrovo
  - Complex Oncology Center Rousse Eood, Rousse
  - Mhat For Womens Health Nadezhda, Ood, Sofia
  - Acibadem City Clinic Mhat Tokuda Ead, Sofia
- China (44):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital Branch North, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Province Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Union Medical Center (Nankai University Affiliated Hospital), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics Branch Oncology Hospital, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - National Cancer Institute, Vilnius
- Mexico (7):
  - Investigacion Onco Farmaceutica (Oncotech), La Paz
  - Fundacion Rodolfo Padilla Padilla, Ac, León
  - Health Pharma Professional Research Sa de Cv, Mexico City
  - Medica Sur, México
  - Accelerium S de Rl de Cv, Monterrey
  - Centro de Investigacion Clinica Chapultepec Sa de Cv, Morelia
  - Oaxaca Site Management Organization Sc, Oaxaca City
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton Waikato
  - Tauranga Hospital, Tauranga
- Poland (9):
  - Szpital Specjalistyczny Brzeziny, Brzeziny
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Terapii Wspolczesnej Jm Jasnorzewska Sp Komandytowo Akcyjna, Lodz
  - Salve Medica Sp Z Oo, Sp Komandytowa, Lodz
  - Zespol Gruzlicy I Chorob Pluc W Olsztynie Oddz Onkologii Z Pododdz Chemioterapii Nowotworow Puc, Olsztyn
  - Mazowiecki Szpital Specjalistyczny W Ostrolece Im Dr Jozefa Psarskiego, Ostrołęka
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy, Otwock
  - Izerskie Centrum Pulmonologii I Chemioterapii Izer Med Spolka Z Oo, Szklarska Porba
  - Centrum Onkologii Instytut Im M Sklodowskiej Curie, Warsaw
- Russia (14):
  - Arkhangelsk Regional Clinical Oncological Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - Irkutsk Regional Oncology Dispensary, Irkutsk, Irkutiskaya Oblast'
  - Fsbi of Higher Educationogarev Mordovia State University, Saransk, Mordoviya, Respublika
  - N N Blokhin Russian Cancer Research Center Konstantin Laktionov, Moscow, Moscow
  - Fsbi Russian Scientific Center of Radiology and Nuclear Medicine of the Moh of the Rf, Moscow, Moscow
  - Vitamed Llc, Moscow, Moscow
  - Bih of Omsk Region Clinical Oncology Dispensary, Omsk, Omsk Oblast
  - Sbei Hpe Ryazan State Medical University Na Academician Ip Pavlov of the Moh of the Rf, Ryazan, Ryazan Oblast
  - Private Medical Institution Evromedservis, Pushkin, Sankt-Peterburg
  - Pavlov First Saint Petersburg State Medical University, SaintPetersburg, Sankt-Peterburg
  - Llc Center of Palliative Medicine Devita, SaintPetersburg, Sankt-Peterburg
  - Fsbi Clinical Research and Practical Center For Specialized Medical Care (Oncology), SanktPetersburg, Sankt-Peterburg
  - State Budgetary Healthcare Institution Volgograd Regional Clinical Oncology Dispensary, Volgograd, Volgograd Oblast
  - Fsbi National Medical Research Center For Oncology Na Nn Petrov of the Moh of the Rf, SaintPetersburg
- Slovakia (8):
  - Fakultna Nemocnica S Poliklinikou Fd Roosevelta, Banská Bystrica
  - Nemocnica S Poliklinikou Sv Jakuba, No Bardejov, Bardejov
  - Narodny Onkologicky Ustav, Bratislava
  - Vychodoslovensky Onkologicky Ustav, As, Košice
  - Nemocnica S Poliklinikou Stefana Kukuru Michalovce, As, Michalovce
  - Fakultna Nemocnica S Poliklinikou Nove Zamky, Nové Zámky
  - Nemocnica Na Okraji Mesta, No, Partizánske
  - Poko Poprad Sro, Poprad
- Turkey (Türkiye) (11):
  - Acibadem Adana Hospital, Adana
  - Hacettepe University, Ankara
  - Nonu Universitesi Tip Fakultesi, Battalgazi
  - Tr Trakya University Health Research and Application Center (Hospital), Edirne
  - Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Ehir Hastanesi, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Necmettin Erbakan University Selcuklu Faculty of Medicine, Meram
  - Iu C, Clinical Research Excellence Application and Research Center, Stanbul
  - Namik Kemal University, Tekirdağ

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Zhou C, Huang D, Fan Y, Yu X, Liu Y, Shu Y, Ma Z, Wang Z, Cheng Y, Wang J, Hu S, Liu Z, Poddubskaya E, Disel U, Akopov A, Dvorkin M, Zheng W, Ma Y, Wang Y, Li S, Yu C, Rivalland G. Tislelizumab Versus Docetaxel in Patients With Previously Treated Advanced NSCLC (RATIONALE-303): A Phase 3, Open-Label, Randomized Controlled Trial. J Thorac Oncol. 2023 Jan;18(1):93-105. doi: 10.1016/j.jtho.2022.09.217. Epub 2022 Sep 29. PMID 36184068
- [Result] Huang D, Zhou C, Barnes G, Ma Y, Li S, Zhan L, Tang B. The effects of tislelizumab treatment on the health-related quality of life of patients with advanced non-small cell lung cancer. Cancer Med. 2023 Aug;12(16):17403-17412. doi: 10.1002/cam4.6361. Epub 2023 Aug 17. PMID 37587845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 109 study centers in 10 countries (China, Brazil, Bulgaria, Lithuania, Mexico, New Zealand, Poland, Russia, Slovakia, and Turkey).
Pre-assignment Details: Eligible participants were randomized in a 2:1 ratio to receive either tislelizumab or docetaxel treatment. Randomization was stratified by histology (squamous versus non--squamous), line of therapy (second line versus third line), and programmed cell death protein ligand-1 (PD-L1) expression (≥ 25% tumor cells (TCs) versus < 25% TCs).
Period: Overall Study
Arm/Group | Tislelizumab | Docetaxel
Started | 535 | 270
Received Treatment | 534 | 258
Completed | 0 | 0
Not Completed | 535 | 270
Not completed — Death | 409 | 223
Not completed — Study Closed by Sponsor | 66 | 29
Not completed — Withdrawal by Subject | 13 | 16
Not completed — Lost to Follow-up | 13 | 2
Not completed — Miscellaneous | 33 | 0
Not completed — Remained on Study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tislelizumab: Participants received tislelizumab 200 mg IV once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of informed consent, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Tislelizumab | Docetaxel | Total
Number analyzed (Participants) | 535 | 270 | 805
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.79) | 60.7 (8.95) | 60.5 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 64 | 183
  Male | 416 | 206 | 622
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 1 | 13
  Asian | 424 | 219 | 643
  Black or African American | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  White | 93 | 44 | 137
  Other | 2 | 0 | 2
Histology [Count of Participants; unit: Participants]
  Squamous | 248 | 122 | 370
  Non-Squamous | 287 | 148 | 435
Current Line of Therapy [Count of Participants; unit: Participants]
  Second line | 453 | 229 | 682
  Third line | 82 | 41 | 123
PD-L1 Expression [Count of Participants; unit: Participants] — Participants were tested for PD-L1 expression by a central laboratory using VENTANA SP263 immunohistochemistry assay.
  Participants
    ≥ 25% of tumor cells | 227 | 115 | 342
    < 25% of tumor cells | 307 | 152 | 459
    Missing | 1 | 3 | 4
Smoking Status [Count of Participants; unit: Participants]
  Never | 162 | 82 | 244
  Current | 50 | 20 | 70
  Former | 323 | 168 | 491

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in All Participants (Co-primary Endpoint)
Description: OS was defined as the time from randomization to death from any cause. Median OS was calculated using the Kaplan-Meier method. Data for participants who were not reported as having died at the time of analysis were censored at the date they were last known to be alive. Data for participants who did not have postbaseline information were censored at the date of randomization.
Time Frame: From randomization to the data cutoff date of 10 August 2020; up to 32.4 months
Population: The Intent-to-Treat (ITT) Analysis Set included all randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 535 | 270
months | 17.2 [15.28 to 20.04] | 11.9 [10.18 to 13.93]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; Test type: Superiority; p < 0.0001, 1-sided Log Rank Test — OS in the ITT population was tested at one-sided p value boundary of 0.0120; Stratified by stratification factors: histology (squamous vs non-squamous), line of therapy (second vs third), and PDL1 expression (≥25% vs <25% TC); Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.527 to 0.778] — A stratified Cox proportional hazards model with Efron's method of tie handling was used to determine hazard ratio (HR) and its 95% confidence interval (CI)

2. Primary Outcome: Overall Survival (OS) in Programmed Cell Death Protein Ligand-1 (PD-L1)-Positive Participants (Co-primary Endpoint)
Description: as for outcome 1
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 15 July 2021; Up to 43 months
Population: The PD-L1-Positive Analysis Set included all randomized patients whose tumors were PD-L1 positive (defined as ≥ 25% of tumor cells with PD-L1 membrane staining).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 227 | 115
months | 19.3 [16.49 to 22.60] | 11.5 [8.15 to 13.54]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; Test type: Superiority; p < 0.0001, 1-sided Log Rank Test — OS in the PD-L1 positive analysis set was tested at the one-sided p-value boundary of 0.025; Stratified by stratification factors: histology (squamous vs non-squamous) and line of therapy (second vs third); Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.407 to 0.702]

3. Secondary Outcome: Objective Response Rate (ORR) in All Participants
Description: Objective response rate is defined as the percentage of participants who had a complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 Tumor assessments included computed tomography (CT) scans or magnetic resonance imaging (MRI), with preference for CT, of the chest, abdomen, and pelvis.
  CR: Disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the size of target lesions and no progression of non-target lesions and no new lesions, or disappearance of all target lesions with persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits and no new lesions.
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 15 July 2021; Up to 43 months
Population: Intent-to-Treat Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 535 | 270
percentage of participants | 22.6 [19.14 to 26.40] | 7.0 [4.29 to 10.77]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) chi-square test stratified by histology, line of therapy, and PDL1 expression; Odds Ratio (OR) = 3.86, 95% CI 2-sided [2.336 to 6.393]

4. Secondary Outcome: Objective Response Rate in PD-L1-Positive Participants
Description: as for outcome 3
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 15 July 2021; Up to 43 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 227 | 115
percentage of participants | 37.4 [31.13 to 44.09] | 7.0 [3.05 to 13.25]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) chi-square test stratified by histology and line of therapy; Odds Ratio (OR) = 8.04, 95% CI 2-sided [3.721 to 17.379]

5. Secondary Outcome: Duration of Response (DOR) for All Responders
Description: DoR was defined as the time from the first documented objective response to documented disease progression as assessed by the investigator using RECIST v1.1, or death from any cause, whichever occurred first.
  Median DOR was estimated using the Kaplan-Meier method.
  Progressive Disease (PD): At least a 20% increase in the size of target lesions with an absolute increase of at least 5 mm, or unequivocal progression of existing non-target lesions, or the appearance of any new lesions.
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 15 July 2021; Up to 43 months
Population: Participants in the Intent-to-Treat Analysis Set who had an objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 121 | 19
months | 13.5 [8.54 to 19.58] | 6.0 [2.10 to 7.16]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; Test type: Superiority; p < 0.0001, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.176 to 0.536] — A stratified Cox proportional hazards model with Efron's method of tie handling was used to determine hazard ratio (HR) and its 95% CI

6. Secondary Outcome: Duration of Response (DOR) in PD-L1-Positive Responders
Description: as for outcome 5
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 15 July 2021; Up to 43 months
Population: Participants in the PD-L1-Positive Analysis Set who had an objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 85 | 8
months | 11.9 [8.31 to 19.58] | 4.2 [0.56 to 6.05]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; Test type: Superiority; p < 0.0001, Log Rank; Stratified by stratification factors: histology (squamous vs non-squamous) and line of therapy (second vs third); Hazard Ratio (HR) = 0.16, 95% CI 2-sided [0.066 to 0.370] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Progression-free Survival (PFS) in All Participants
Description: PFS was defined as the time from randomization to the first objectively documented disease progression as assessed by the investigator per RECIST v1.1 or death from any cause, whichever occurred first.
  Median PFS was estimated using the Kaplan-Meier method.
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 15 July 2021; Up to 43 months
Population: Intent-to-Treat Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 535 | 270
months | 4.2 [3.88 to 5.52] | 2.6 [2.17 to 3.78]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; Test type: Superiority; p < 0.0001, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.528 to 0.745] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Progression-free Survival in PD-L1 Positive Participants
Description: as for outcome 7
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 15 July 2021; Up to 43 months
Population: PD-L1 Positive Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 227 | 115
months | 6.5 [6.24 to 8.28] | 2.5 [2.10 to 4.11]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; Test type: Superiority; p < 0.0001, Log Rank; Stratified by stratification factors: histology (squamous vs non-squamous) and line of therapy (second vs third); Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.285 to 0.494] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (GHS)/Quality of Life (QOL) Score
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and two global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. Higher scores in GHS/QoL score indicates better quality of life.
Time Frame: Baseline and Cycle 6 (each cycle was 3 weeks)
Population: The HRQoL Analysis Set included all randomized participants who received ≥ 1 dose of study drug and completed ≥ 1 HRQoL assessment; participants with available data at baseline and Cycle 6 are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 316 | 76
score on a scale | 2.4 [0.62 to 4.12] | -3.4 [-6.45 to -0.27]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; The linear mixed-effect model for repeated measures (MMRM) includes baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects and visit as a repeated measure; Test type: Other; p = 0.0008, Mixed Models Analysis; Least Squares (LS) Mean Difference = 5.7, 95% CI 2-sided [2.38 to 9.07]

10. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire Lung Cancer 13 Items (QLQ-LC13) Coughing, Dyspnoea, and Chest Pain Scores
Description: The EORTC QLQ-LC13 is the lung cancer module of the QLQ-C30 and measures lung cancer-specific disease and treatment symptoms. It includes 13 questions about specific symptoms in which participants respond based on a 4-point scale, where 1 is "not at all" and 4 is "very much". Raw scores are transformed into a 0 to 100 scale via linear transformation. Lower scores indicate an improvement in symptoms.
Time Frame: Baseline and Cycle 6 (each cycle was 3 weeks)
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 316 | 77
score on a scale
  Coughing Scale | -7.8 [-10.23 to -5.30] | 0.5 [-3.87 to 4.87]
  Dyspnoea Scale | -1.2 [-2.93 to 0.56] | 2.0 [-1.01 to 5.05]
  Chest Pain Scale | -0.9 [-2.86 to 1.06] | 1.3 [-2.15 to 4.84]
Statistical Analysis 1: Comparison: Tislelizumab vs Docetaxel; Analysis of Change from Baseline in Coughing Scale. The linear mixed-effect model for repeated measures (MMRM) includes baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects and visit as a repeated measure; Test type: Other; p = 0.0007, Mixed Models Analysis; LS Mean Difference = -8.3, 95% CI 2-sided [-13.02 to -3.51]
Statistical Analysis 2: Comparison: Tislelizumab vs Docetaxel; Analysis of Change from Baseline in Dyspnoea Scale. The linear mixed-effect model for repeated measures (MMRM) includes baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects and visit as a repeated measure; Test type: Other; p = 0.0579, Mixed Models Analysis; LS Mean Difference = -3.2, 95% CI 2-sided [-6.52 to 0.11]
Statistical Analysis 3: Comparison: Tislelizumab vs Docetaxel; Analysis of Change from Baseline in Chest Pain Scale. The linear mixed-effect model for repeated measures (MMRM) includes baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects and visit as a repeated measure; Test type: Other; p = 0.2472, Mixed Models Analysis; LS Mean Difference = -2.2, 95% CI 2-sided [-6.05 to 1.56]

11. Secondary Outcome: Change From Baseline in European Quality of Life 5-Dimensions, 5-level (EQ-5D-5L) Visual Analogue Scale (VAS)
Description: The EQ-5D-5L measures health outcomes using a VAS to record a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine.' A higher score indicates better health outcomes.
Time Frame: Baseline and Cycle 6 (each cycle was 3 weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 237 | 60
score on a scale | 1.0 (11.89) | 1.7 (11.36)

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered related to study drug or not.
  The investigator assessed the severity of each AE and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03 as defined below:
  * Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  * Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate activities of daily living.
  * Grade 3: Severe or medically significant but not immediately life threatening. hospitalization or prolongation of hospitalization indicated; disabling; limiting selfcare activities of daily living.
  * Grade 4: Life threatening consequences; urgent intervention indicated.
  * Grade 5: Death related to AE.
Time Frame: From first dose of study drug to 30 days after last dose, up to the study completion date cut-off date of 18 January 2024 (up to approximately 63 months)
Population: The Safety Analysis Set included all randomized patients who received ≥ 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tislelizumab | Docetaxel
Number analyzed (Participants) | 534 | 258
Participants
  Any TEAE | 518 | 254
  ≥ Grade 3 TEAE | 233 | 193

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from randomization up to study completion date cut-off date of 18 January 2024, up to 63 months. AEs are reported from first dose of study drug to 30 days after last dose, up to study completion date cut-off date of 18 January 2024, up to 63 months.
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events includes all randomized participants who received ≥ 1 dose of any study treatment.
Arm/Group | Tislelizumab | Docetaxel
All-Cause Mortality (participants affected / at risk) | 409/535 | 223/270
Serious Adverse Events (participants affected / at risk) | 192/534 | 84/258
Other Adverse Events (participants affected / at risk) | 498/534 | 246/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=534) | Docetaxel (N=258)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 21 (22)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 6 (7)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 11 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 5 (5) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Immune-mediated adrenal insuficiency (Endocrine disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 6 (6) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 39 (48) | 19 (21)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Cerebral radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 8 (10)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (5) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Visual pathway disorder (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=534) | Docetaxel (N=258)
Anaemia (Blood and lymphatic system disorders) | 156 (269) | 114 (169)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 13 (13)
Leukopenia (Blood and lymphatic system disorders) | 17 (38) | 70 (169)
Neutropenia (Blood and lymphatic system disorders) | 10 (24) | 73 (185)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (28) | 9 (22)
Hyperthyroidism (Endocrine disorders) | 23 (23) | 0 (0)
Hypothyroidism (Endocrine disorders) | 66 (82) | 2 (2)
Cataract (Eye disorders) | 22 (23) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 8 (8) | 12 (14)
Abdominal pain upper (Gastrointestinal disorders) | 16 (20) | 10 (11)
Constipation (Gastrointestinal disorders) | 74 (89) | 44 (51)
Diarrhoea (Gastrointestinal disorders) | 41 (52) | 35 (51)
Nausea (Gastrointestinal disorders) | 65 (73) | 43 (55)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 12 (14)
Toothache (Gastrointestinal disorders) | 20 (23) | 6 (7)
Vomiting (Gastrointestinal disorders) | 35 (44) | 19 (23)
Asthenia (General disorders) | 76 (78) | 57 (64)
Chest discomfort (General disorders) | 19 (19) | 8 (8)
Chest pain (General disorders) | 21 (21) | 2 (2)
Fatigue (General disorders) | 37 (40) | 24 (31)
Malaise (General disorders) | 40 (44) | 17 (28)
Non-cardiac chest pain (General disorders) | 22 (29) | 7 (9)
Oedema peripheral (General disorders) | 15 (15) | 10 (11)
Pyrexia (General disorders) | 62 (72) | 26 (29)
Pneumonia (Infections and infestations) | 40 (43) | 18 (19)
Upper respiratory tract infection (Infections and infestations) | 55 (76) | 23 (25)
Alanine aminotransferase increased (Investigations) | 112 (183) | 39 (47)
Aspartate aminotransferase increased (Investigations) | 106 (172) | 32 (38)
Bilirubin conjugated increased (Investigations) | 17 (25) | 7 (9)
Blood alkaline phosphatase increased (Investigations) | 39 (53) | 10 (13)
Blood bilirubin increased (Investigations) | 36 (49) | 15 (23)
Blood creatine phosphokinase MB increased (Investigations) | 21 (34) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 47 (97) | 2 (4)
Blood creatinine increased (Investigations) | 37 (58) | 17 (22)
Blood lactate dehydrogenase increased (Investigations) | 38 (48) | 18 (23)
Blood thyroid stimulating hormone increased (Investigations) | 32 (56) | 3 (3)
Blood urea increased (Investigations) | 26 (38) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 31 (47) | 15 (19)
Lymphocyte count decreased (Investigations) | 35 (76) | 18 (37)
Neutrophil count decreased (Investigations) | 17 (38) | 90 (168)
Neutrophil count increased (Investigations) | 19 (23) | 7 (9)
Platelet count decreased (Investigations) | 21 (37) | 9 (11)
Weight decreased (Investigations) | 90 (101) | 31 (32)
White blood cell count decreased (Investigations) | 21 (58) | 75 (133)
White blood cell count increased (Investigations) | 20 (30) | 11 (13)
Decreased appetite (Metabolism and nutrition disorders) | 88 (95) | 62 (71)
Hyperglycaemia (Metabolism and nutrition disorders) | 56 (111) | 29 (37)
Hyperuricaemia (Metabolism and nutrition disorders) | 24 (52) | 7 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 76 (141) | 40 (64)
Hypocalcaemia (Metabolism and nutrition disorders) | 29 (49) | 21 (26)
Hypochloraemia (Metabolism and nutrition disorders) | 19 (29) | 11 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 51 (83) | 14 (16)
Hyponatraemia (Metabolism and nutrition disorders) | 53 (85) | 28 (37)
Hypophosphataemia (Metabolism and nutrition disorders) | 11 (25) | 9 (16)
Hypoproteinaemia (Metabolism and nutrition disorders) | 22 (27) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 68 (83) | 23 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 41 (47) | 20 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 16 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 (36) | 17 (23)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (25) | 8 (9)
Dizziness (Nervous system disorders) | 19 (21) | 13 (15)
Headache (Nervous system disorders) | 23 (28) | 12 (12)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 13 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 9 (10)
Insomnia (Psychiatric disorders) | 34 (58) | 26 (29)
Proteinuria (Renal and urinary disorders) | 17 (26) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 111 (128) | 40 (46)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62 (64) | 31 (35)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 51 (62) | 17 (18)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 36 (49) | 22 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 127 (130)
Pruritus (Skin and subcutaneous tissue disorders) | 41 (44) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 38 (41) | 7 (7)
Hypertension (Vascular disorders) | 25 (32) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT03358875/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT03358875/SAP_001.pdf